CLINICAL TRIAL: NCT04427813
Title: Sexual and Marital Health and Problems During the Covid -19 in the Last Months
Brief Title: Sexual Health and Problems During the Covid -19 Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher , lecturer ,Obstetrics and Gynecology , National Research Centre, Aljazeera Hospital
Other Study IDs: marital health
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Sexual Behavior
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionaire to husband and wife — a form of questions will be asked to every partner

SUMMARY:
Covid-19 is an emerging critical highly infectious virus

DETAILED DESCRIPTION:
The covid-19 pandemic is a very harmful crisis that affects all human activities

ELIGIBILITY:
Inclusion Criteria:

* any partners between 18-60 years

Exclusion Criteria:

* any husband or wife that have organic sexual problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: partners betwen 18-60 years
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-06-11 (Estimated); Primary Completion 2020-07-05 (Estimated); Study Completion 2020-07-12 (Estimated)

PRIMARY OUTCOMES:
the number of partners that have unusual behaviour | One month
  the husband and wife who have abnormal behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt